CLINICAL TRIAL: NCT04707755
Title: Effects of Motor Imagery Technique on Lower Limb Function Among Stroke Patients.
Brief Title: Motor Imagery Technique on Lower Limb Function Among Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC00664 Izharuddin
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Spasticity as Sequela of Stroke; Gait, Hemiplegic; Quality of Life
Keywords: Gait; Lower Limb function; Motor imagery
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor imagery technique (Experimental): Motor Imagery technique Plus Conventional Physical therapy
  Interventions: Other: Motor imagery technique
- Conventional Physical therapy (Active Comparator): passive stretching, ROM exercises, sitting to standing, anteroposterior step, climbing and descending stairs.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Motor imagery technique — The patient will sit on chair in a quiet room. The patients will be observing motor performance in video, motor performance video will consist of (1) knee flexion and extension movement, (2) sitting to standing movement, (3) stepping movement, (4) walking, (5) climbing and descending stairs.
  Addition to motor imagery, the patients will be provided the passive stretching, ROM exercises, sitting to standing, anteroposterior step, climbing and descending stairs.
  Arms: Motor imagery technique
Other: Conventional Physical Therapy — It includes passive stretching, ROM exercises, sitting to standing, anteroposterior step, climbing and descending stairs.
  Arms: Conventional Physical therapy

SUMMARY:
To determine the effects of motor imagery technique on lower limb function among stroke patient.

To determine the effects of motor imagery technique on lower limb spasticity among stroke patients.

To determine the effects of motor imagery technique on gait among stroke patients.

To determine the effects of motor imagery technique on quality of life among stroke patients

DETAILED DESCRIPTION:
Stroke affected the functional capacities and the state of health thus altered quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult without ADHD by Adult ADHD Self-Report Scale score.
* History of no more than one stroke.
* Lower limb muscles spasticity with the grade 1+ or 2 on modified Ashworth in scale.
* Mini-mental status score more than 25.
* Patients who are less than 6 months post-stroke.
* Modified Rankin scale score is 4.

Exclusion Criteria:

* Lesion of frontal, parietal and basal ganglia
* Excessive spasticity that is score of>3 on modified Ashworth spasticity scale.
* Any musculoskeletal disorder impeding lower limb function.
* Participating in any experimental rehabilitation or drug studies.
* Bed ridden patient.
* Subjects psychiatric disorder or dementia.
* Any neglect of space on the affected side, or any other neurological disease or auditory or visual.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Function scale | 8 weeks
  It is 20 items questionnaire, measure the lower extremity function scoring from 1 to 4 for each items, in which minimum score is 0 and maximum score of 80 shows the maximum functional status. It has a valid and reliable tool to measure the lower extremity functional status.
Dynamic Gait Index | 8 weeks
  It assess gait, balance and fall risk, with 24 is the maximum score, in which 19 or less have been related to increase incidence of falls. It has high reliability and validity in the stroke population.
Time Up and Go test | 8 weeks
  It assess a person's mobility and requires both static and dynamic balance. Score of less than 10 seconds indicate freely mobile,<20 seconds mostly independent, 20-29 seconds variable mobility, >30 seconds Impaired mobility. It is reliable, valid, and easy to administer clinical tool in stroke patients.
Stroke Specific Quality of Life Scale | 8 Weeks
  It is a self-report questionnaire, measure the quality of life in stroke patients consisting of 49 items in the 12 domains. Scoring from 1 to 5 , in which 1 shows strongly agreement and 5 shows strongly disagreement. It is a reliable and valid tool for measuring the quality of life for stroke patients.
Modified Ashworth scale | 8 Weeks
  It measures the spasticity, ranging from 0 means normal tone to 4 shows increased tone to such extent where passive movement is not possible. It has good intra-rater reliability and validity in stroke patients .

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- Bibi Zahida Memorial Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gul I, Malik MS, Halim A, Rauf S. POST STROKE DEPRESSION: EXPERIENCE AT A TERTIARY CARE HOSPITAL OF PAKISTAN. Pakistan Armed Forces Medical Journal. 2019 Aug 27;69(4):779-83.
- [Background] Paravlic AH, Pisot R, Marusic U. Specific and general adaptations following motor imagery practice focused on muscle strength in total knee arthroplasty rehabilitation: A randomized controlled trial. PLoS One. 2019 Aug 14;14(8):e0221089. doi: 10.1371/journal.pone.0221089. eCollection 2019. PMID 31412056
- [Background] Pedersen SG, Heiberg GA, Nielsen JF, Friborg O, Stabel HH, Anke A, Arntzen C. Validity, reliability and Norwegian adaptation of the Stroke-Specific Quality of Life (SS-QOL) scale. SAGE Open Med. 2018 Jan 8;6:2050312117752031. doi: 10.1177/2050312117752031. eCollection 2018. PMID 29344360